CLINICAL TRIAL: NCT02285023
Title: Cross-Cultural of the Validity, Reliability and Interpretability of Thai-version of Chronic Urticaria Quality of Life Questionnaire (CU-Q2oL)
Brief Title: The Validity, Reliability and Interpretability of Thai-version of Chronic Urticaria Quality of Life Questionnaire
Acronym: CU-Q2oL
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Collaborators: University of Genua, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: Thai-version of CU-Q2oL
Record Dates: First submitted 2014-10-17; First posted 2014-11-06 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2018-09

CONDITIONS: Chronic Urticaria
Keywords: Chronic urticaria; CU-Q2oL
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CU-Q2oL: * Evaluation by the Urticaria Activity Score (UAS7)
  * Fill the DLQI and CU-Q2oL questionnaire
  Interventions: Other: CU-Q2oL

INTERVENTIONS:
Other: CU-Q2oL — The patients will be explained how to complete the Urticaria Activity Score (UAS7) form for evaluating their severity of chronic urticaria symptoms at home.
  At the 2nd visit, collect the 1st UAS7 assessment. Assessment the severity of chronic urticaria symptoms. The patients fill the 1st DLQI and CU-Q2oL questionnaire and get the 2nd UAS7 form and two-week appointment to follow up.
  At the 3th visit, collect the 2nd UAS7 assessment. Assessment the severity of chronic urticaria symptoms. The patients fill the 2nd DLQI and CU-Q2oL questionnaire.

SUMMARY:
In the majority of patients with the chronic urticaria, the etiology is unclear, leading to difficulties in treatment and high rates of recurrence. According to the International EAACI/GA2LEN/EDF/WAO Guidelines (the Dermatology Section of the European Academy of Allergology and Clinical Immunology(EAACI), the Global Allergy and Asthma European Network (GA2LEN), the European Dermatology Forum (EDF) and the World Allergy Organization (WAO) in Urticaria, using the Chronic Urticaria Quality of Life Questionnaire in a routine management is the key for a better treatment outcome. To translate this questionnaire into Thai is essential in our subject of interest in order to effectively apply it to local patients. The Thai-version questionnaire will encourage enhanced as well as impactful therapeutic options for Thai chronic urticaria patients.

DETAILED DESCRIPTION:
1. Adaption of the Cu-Q2oL questionnaire into Thai version by using forward-backward translation that is independently performed by two bilingual translators. The original Italian version is translated into Thai by two Thai native speakers, then the study team reviews the Thai-version Cu-Q2oL questionnaire for items comprehensibility and integrates the first consensus version which re-translated into Italian by an Italian native speaker afterwards. The comparison between the backward Italian version Cu-Q2oL questionnaire and the original Cu-Q2oL is carried out to find out whether there are any misconception and mistranslation in the intermediary forward version of questionnaire. After that, the second consensus version will be tested on 15 chronic urticaria patients to detect any misunderstanding points based on patients' comments. Finally, this Thai-version of CU-Q2oL questionnaire will be used to investigate the validity, reliability, interpretability and minimal clinical important difference.
2. To investigate the validity, reliability and interpretability of Thai-version of Chronic Urticaria Quality of Life Questionaire (CU-Q2oL), the severity of chronic urticaria symptoms will be assessed by investigators and patients using the Urticaria Activity Score (UAS7), the DLQI and CU-Q2oL questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or above
* Diagnosed as chronic urticaria based on "The EAACI/GA(2)LEN/EDF/WAO Guideline
* Literate in Thai language and can complete the questionnaire by themselves

Exclusion Criteria:

* Have other active skin diseases
* Have a psychiatric problem
* Cannot understand the questionnaire by themselves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were diagnosed as chronic urticaria.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2014-11; Primary Completion 2015-02 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kanokwalai Kulthanan, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients diagnosed as chronic idiopathic urticaria were invited to participate in the study at the Allergy clinic in the Department of Dermatology, Siriraj Hospital, Mahidol University, Bangkok, Thailand.
Groups:
- CU-Q2oL: * Evaluation by the Urticaria Activity Score (UAS7)
  * Fill the DLQI and CU-Q2oL questionnaire
  CU-Q2oL: The patients will be explained how to complete the Urticaria Activity Score (UAS7) form for evaluating their severity of chronic urticaria symptoms at home.
  At the 2nd visit, collect the 1st UAS7 assessment. Assessment the severity of chronic urticaria symptoms. The patients fill the 1st DLQI and CU-Q2oL questionnaire and get the 2nd UAS7 form and two-week appointment to follow up.
  At the 3th visit, collect the 2nd UAS7 assessment. Assessment the severity of chronic urticaria symptoms. The patients fill the 2nd DLQI and CU-Q2oL questionnaire.
Period: Overall Study
Arm/Group | CU-Q2oL
Started | 166
Completed | 166
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients diagnosed as chronic idiopathic urticarial were enrolled.
Groups:
- Chronic Idiopathic Urticaria Patients: * Evaluation by the Urticaria Activity Score (UAS7)
  * Fill the DLQI and CU-Q2oL questionnaire
  CU-Q2oL: The patients diagnosed as chronic idiopathic urticaria will be explained how to complete the Urticaria Activity Score (UAS7) form for evaluating their severity of chronic urticaria symptoms at home.
  At the 2nd visit, collect the 1st UAS7 assessment. Assessment the severity of chronic urticaria symptoms. The patients fill the 1st DLQI and CU-Q2oL questionnaire and get the 2nd UAS7 form and two-week appointment to follow up.
  At the 3th visit, collect the 2nd UAS7 assessment. Assessment the severity of chronic urticaria symptoms. The patients fill the 2nd DLQI and CU-Q2oL questionnaire.
Arm/Group | Chronic Idiopathic Urticaria Patients
Number analyzed (Participants) | 166
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 166
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131
  Male | 35
Region of Enrollment [Number; unit: participants]
  Thailand | 166
Urticaria Activity Score [Mean (Standard Deviation); unit: units on a scale] — The UAS is a specific questionnaire to determine the disease severity of CU patients over one week (UAS7). The UAS7 represents daily numbers of wheals (range: 0-none to 3-severe) and severity of pruritus (range: 0-none to 3-severe) for the 7 days with the maximum sum score of 42.15 The severity is classified as follows: severe (28-42), moderate (16-27), mild (7-15), well-controlled (1-6), and complete response (0). The UAS7 scores were recorded by the patient themselves seven days prior to each visit.
  units on a scale | 8.8 (9.6)
Dermatology Life Quality Index [Mean (Standard Deviation); unit: Score] — The DLQI is an HRQoL questionnaire for general dermatologic diseases that was developed by Finlay and Khan. It comprises 10 questions corresponding to six domains: Symptoms and feeling, Daily activities, Leisure, Work and school, Personal relationships, and Treatment. The total DLQI score ranges from 0 to 30. Dr. Finlay previously gave formal permission to the first author to validate and use the Thai version of the DLQI questionnaire. The DLQI Scores of 0-1, 2-5, 6-10, 11-20, and 21-30 mean no effect, small effect, moderate effect, very large effect, extremely large effect on quality of life.
  Score | 4.67 (5.3)
CU-Q2OL [Mean (Standard Deviation); unit: units on a scale] — The Thai version of the CU-Q2oL questionnaire comprises 23 items categorized into three domains: domain I (sleep, leisure, concentration) domain II (symptomatic, eating limits), domain III (mental status, looks, impact on life activities). For each item, patients were asked to choose between five response values (scored 0-4) indicating the intensity of each item in the last 2 weeks. A total summed score across all items was calculated and transformed into scores ranging from 0 to 100, with a score of 100 indicating the worst HRQoL impairment.
  units on a scale | 19.91 (15.9)
Education [Number; unit: participants] — Participants completing at least primary school education
  participants | 166

OUTCOME MEASURES:

1. Primary Outcome: Cross-Cultural Validity of Thai-version CU-Q2oL
Description: Cross-cultural validity is the degree to which the performance of the Thai CU-Q2oL items can adequately reflect the performance of the original CU-Q2oL items. Exploratory factor analysis was used to determine scales with proper item division of the Thai CU-Q2oL. Principal component analysis with varimax rotation was employed. An eigenvalue ≥ 1 was chosen as the criterion to retain domains. Each item was classified into the domain when loading with a domain loading ≥ 0.5.
Time Frame: 4 week
Measure: Number; unit: Percentage
Groups:
- Extraction Sums of Square Loading (% of Variance): % of Variance - This column contains the percent of total variance accounted for by each factor.
- Rotation Sums of Squared Loading (% of Variance): The "% of variance" column tells you how much of the total variability (in all of the variables together) can be accounted for by each of these summary scales or factors.
Arm/Group | Extraction Sums of Square Loading (% of Variance) | Rotation Sums of Squared Loading (% of Variance)
Number analyzed (Participants) | 166 | 166
Percentage
  Domain I (item 7,8,11-14 of CUQoL) | 43.71 | 22.11
  Domain II( Item 1-6, 9-10, 17 of CUQoL) | 9.41 | 20.21
  Domain III (Item 15-16, 18-23 of CUQoL) | 7.33 | 18.13
Statistical Analysis 1: Comparison: Extraction Sums of Square Loading (% of Variance) vs Rotation Sums of Squared Loading (% of Variance); Exploratory factor analysis; Test type: Non-Inferiority or Equivalence — Principal component analysis with varimax rotation was employed. An eigenvalue ≥ 1 was chosen as the criterion to retain domains. Each item was classified into the domain when loading with a domain loading ≥ 0.5; p < 0.01, exploratory factor analysis — An eigenvalue ≥ 1 was chosen as the criterion to retain domains. Each item was classified into the domain when loading with a domain loading ≥ 0.5; An eigenvalue ≥ 1 was chosen as the criterion to retain domains. Each item was classified into the domain when loading with a domain loading ≥ 0.5

2. Secondary Outcome: Mean Total Score and Domain of Thai CU-Q2oL Scores From the Thai Version to Investigate Reliability of Thai-Version CU-Q2oL
Description: - The CU-Q2oL Questionnaire is a 23-item HRQoL questionnaire. It measures three dimensions (scales) of HRQoL: domain I (sleep, leisure, concentration), domain II (symptom, eating limits), and domain III (mental status, looks, impact on life activities) The scores of domain I of CUQ2oL range between 0 and 26. The scores of domain II of CUQ2oL range between 0 and 39.The scores of domain III of CUQ2oL between 0 and 35.
  The minimum possible score is 0 and the maximum possible score is 100 for total scale.
  -The DLQI scores range from 0-30. Domain I (leisure), Domain II (symptoms and feeling), and Domain III (daily activities, work, school, and personal relationships). Meaning of DLQI Scores: 0-1 = no effect, 2-5 = small effect, 6-10 = moderate effect, 11-20 = very large effect, 21-30 = extremely large effect.
  The higher the score, the more quality of life is impaired for both the CUQ2oL and the DLQI.
Time Frame: baseline
Population: Mean score of domain I, II, III of Thai CU-Q2oL were correlated to mean score domain I, II, III of Thai DLQI, respectively
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Mean Score of Thai CUQ2oL at Baseline: It is the sum of individual scores divided by the number of individuals. Minimum and maximum of total CUQ2oL scores are 0 and 100, respectively.
- Mean Score of Thai DLQI at Baseline: It is the sum of individual scores divided by the number of individuals. Minimum and maximum of total DLQI scores are 0 and 30, respectively.
Arm/Group | Mean Score of Thai CUQ2oL at Baseline | Mean Score of Thai DLQI at Baseline
Number analyzed (Participants) | 166 | 166
units on a scale
  Domain I | 23.19 (21.7) | 1.86 (1.4)
  Domain II | 19.09 (16.6) | 1.79 (1.5)
  Domain III | 18.37 (17.5) | 1.85 (2.5)
Statistical Analysis 1: Comparison: Mean Score of Thai CUQ2oL at Baseline; Test type: Superiority or Other; p < 0.05, Crohbach's alpha; Cronbach's alpha = 0.94

3. Secondary Outcome: Change in Thai CU-Q2oL Scores From Baseline for Responders and Non-Responders
Description: - Investigate the smallest reduction in the Thai CU-Q2oL that patients recognized as a meaningful improvement.
Time Frame: baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: score
Groups:
- Responder (Mean): Mean score of the Thai CU-Q2oL of patients who had reduction in DLQI scores higher or equal to 5 were defined as responders.
- Non-responders (Mean): Mean score of the Thai CU-Q2oL of patients who had reduction in DLQI scores less than 5 were defined as non-responders.
Arm/Group | Responder (Mean) | Non-responders (Mean)
Number analyzed (Participants) | 17 | 54
score | 7.3 (9.4) | 28.4 (15.3)

4. Secondary Outcome: Area Under the Curve for Thai CUQ2oL Scores in the Responder Group
Description: The receiver operating characteristic (ROC) analysis and area under the curve (AUC) are acceptable as the units of measure for assess the ability of a questionnaire to changes in patients' health-related quality of life (HRQoL) impairment over time that represents to responsiveness to change and minimal clinical important difference (MCID).
  The AUC of the ROC analysis of 1, 0.9, 0.8, 0.7 and 0.5 were considered perfect, excellent, good, fair, and no better than chance, respectively.
Time Frame: baseline and 2 weeks
Population: Responder group
Measure: Mean (95% Confidence Interval); unit: probability
Groups:
- Area Under the Curve: Patients who had reduction in DLQI scores higher or equal to 5 were defined as responders.
  Patients who had reduction in DLQI scores less than 5 were defined as non-responders.
Arm/Group | Area Under the Curve
Number analyzed (Participants) | 17
probability | 0.90 [0.84 to 0.97]

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Chronic Idiopathic Urticaria: Patients diagnosed as chronic idiopathic urticarial were enrolled.
Arm/Group | Chronic Idiopathic Urticaria
Serious Adverse Events (participants affected / at risk) | 0/166
Other Adverse Events (participants affected / at risk) | 0/166

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No